CLINICAL TRIAL: NCT05495763
Title: The Ultrasonographic Changes of Intercostal Muscles and Diaphragm in Mechanically Ventilated Preterm Neonates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Noha Saied Ibrahim (Other)
Responsible Party: Sponsor-Investigator, Noha Saied Ibrahim, Resident at Pediatrics hospital ainshams university, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: Noha ibrahim
Record Dates: First submitted 2022-08-09; First posted 2022-08-10 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Device: No

SUMMARY:
Invasive mechanical ventilation induces ventilator induced diaphragmatic dysfunction particularly when used for long time and Intercostal muscles as well contribute to the important work of respiratory movement by expanding the thorax , and determining the thickness of them would be a useful parameter in evaluating respiratory muscle activity.

This study will add the impact of mechanical ventilation on the diaphragm and intercostal muscles in preterm infants using ultrasound.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants from 28-36 weeks gestation
2. In need for invasive mechanical ventilation according to work of breathing, oxygen saturation and blood gases .

Exclusion Criteria:

* 1) Significant congenital anomalies including cardiac, abdominal or respiratory.

  2) Congenital anomalies involving the diaphragm. 3) Phrenic nerve paralysis. 4) Congenital muscular dystrophies. 5) Major upper or lower airway anomalies. 6) Storage diseases.

Ages: 5 Minutes to 28 Days | Sex: All
Age Groups: Child
Study Population: The study will be conducted on neonates admitted to NICU.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
The impact of mechanical ventilation on diaphragm and intercostal muscles using ultrasound | 6 months
  Using Ultrasound to measure Intercostal Muscles thickness and diaphragmatic thickness and excursion for assessing the impact of the mechanical ventilation on muscle power predicting weaning from ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt